CLINICAL TRIAL: NCT01312831
Title: A 60-DAY, Open-label, Randomized Study to Evaluate the Efficacy and Safety of Eligen® B12 OR Intramuscularly Administered B12 in Subjects With Low Serum Cobalamin With a 30 Day Extension to 90 Days of Dosing
Brief Title: Efficacy and Safety Study of Oral Eligen® B12 in Subjects With Low Serum Cobalamin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emisphere Technologies, Inc. (Industry)
Responsible Party: M. Cristina Castelli, Ph.D., Emisphere Technologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMIS-112-C-02
Record Dates: First submitted 2011-03-04; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Vitamin B 12 Deficiency
Keywords: cobalamin; B12; homocysteine; MMA; holotranscobalamin; Eligen
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Eligen® B12 (Experimental): Eligen® B12 1000 μg oral tablet taken in the fasted state as a single tablet with 50 mL water. Each dose self-administered daily, for 90 days, after an overnight fast and 1 hour before the morning meal.
  Interventions: Other: Vitamin B12 (cyanocobalamin)
- IM B12 (Active Comparator): Commercially available 1000 μg cyanocobalamin administered IM as 1 mL from a vial containing 1000 μg/mL drug administered by study personnel, in the research clinic, in the morning, in the fasted state and at least 1 hour prior to the morning meal on study Days 1, 3, 7, 10, 14, 21, 30, 60 and 90.
  Interventions: Other: Vitamin B12 (cyanocobalamin)

INTERVENTIONS:
Other: Vitamin B12 (cyanocobalamin)

SUMMARY:
The purpose of this study is to compare the efficacy and safety profile of a new oral vitamin B12 formulation (Eligen® B12) with intramuscular B12 in restoring normal B12 (cobalamin) concentrations in subjects with low cobalamin levels (<350 pg/mL).

ELIGIBILITY:
Inclusion Criteria:

* Vitamin B12 deficiency defined as serum cobalamin below 350 pg/mL
* Age 60 or older; or age 18 or older with gastrointestinal abnormalities including but not limited to gastrointestinal surgery (e.g. gastrectomy, gastric bypass), ileal resection, gastric atrophy, Celiac disease, Crohn's disease, or prolonged use (>3 months) of proton pump inhibitor drugs, or on a restricted diet (such as vegetarian or vegan).
* General good health, as indicated by lack of significant findings in medical history, physical examination, clinical laboratory tests (chemistry, hematology and urinalysis), vital signs, ECG and normal kidney function as determined by estimated creatinine clearance computed with the Cockcroft and Gault formula

Exclusion Criteria:

* Current treatment from a health care provider to treat vitamin B12 deficiency and/or symptoms;
* Daily use of neutralizing antacids (e.g. Maalox®)
* Inability to ingest oral medication
* Clinically significant laboratory value at screening
* Hypersensitivity or allergic reaction to vitamin B12
* Participation in a clinical research study involving a new chemical entity within 30 days of the first study dose
* Folate levels below the reference range provided by the clinical laboratory.
* Renal insufficiency
* Vitamin B6 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-02; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Serum Cobalamin Normalization | 61 days
  The primary efficacy outcome compares the proportion of subjects in each treatment arm in whom cobalamin levels are normalized (i.e., cobalamin ≥ 350 ng/mL) following 60 days of treatment

SECONDARY OUTCOMES:
Maintenance of B12 Normalization | 91 days
  Maintenance of cobalamin normalization after 90 days of treatment
Time to Normalization | 90 days
  Time to normalization of cobalamin levels
Percent Change from Baseline in Cobalamin Levels After 60 and 90 days of Treatment | 91 days
  Change from baseline is defined as (X-B) where B is the baseline (pre-dose Day 1) measurement of cobalamin (pg/mL) and X is the measurement of cobalamin(pg/mL) at Day 61 or Day 91, as required.
  Percent change from baseline is defined as 100(X-B)/B.
Percent Change from Baseline in Methylmalonic Acid (MMA) Levels After 60 and 90 Days of Treatment | 91 days
  Change from baseline is defined as (X-B) where B is the baseline (pre-dose Day 1) measurement of MMA (ng/mL) and X is the measurement of MMA (ng/mL) at Day 61 or Day 91, as required.
  Percent change from baseline is defined as 100(X-B)/B
Percent Change from Baseline in Homocysteine Levels After 60 and 90 Days of Treatment | 91 days
  Change from baseline is defined as (X-B) where B is the baseline (pre-dose Day 1) measurement of homocysteine (umol/L) and X is the measurement of homocysteine (umol/L) at Day 61 or Day 91, as required.
  Percent change from baseline is defined as 100(X-B)/B
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | 91 days
  The safety and tolerability of Eligen® B12 and intramuscular B12 assessed by physical examination findings, clinical laboratory test results, vital signs, 12-lead ECG results and adverse event reporting.
Holo-trancobalamin (holo-TC) Normalization | 91 days
  The proportion of subjects who achieve normalization of holo-TC levels (≥ 40 pmol/L) on Days 61 and 91 as an exploratory endpoint
Holo-TC and Cobalamin Correlation | 91 days
  Holo-TC levels in relation to cobalamin levels on Days 61 and 91 as an exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Benno Roesch, MD, Principal Investigator — Frontage (formerly ABR), 241 Main Street, Hackensack, NJ 07601 USA; Nancy Allegar, MD, Principal Investigator — Alatae Medical LLC, 390 Amwell Road, Building 5, Hillsborough, NJ 08844 USA; Mitchell K. Spinnell, MD, Principal Investigator — Gastroenterology, 1555 Center Avenue, Fort Lee, NJ 07024 USA; Michael M. Rothkopf, MD, Principal Investigator — South Mountain Medical Consultants, 1500 Pleasant Valley Way, Suite 201, West Orange, NJ 07052 USA; Peter Varunok, MD, Principal Investigator — Gastroenterology Associates, 243 North Road, Suite 304, Poughkeepsie, NY 12601 USA

REFERENCES:
- [Derived] Castelli MC, Friedman K, Sherry J, Brazzillo K, Genoble L, Bhargava P, Riley MG. Comparing the efficacy and tolerability of a new daily oral vitamin B12 formulation and intermittent intramuscular vitamin B12 in normalizing low cobalamin levels: a randomized, open-label, parallel-group study. Clin Ther. 2011 Mar;33(3):358-371.e2. doi: 10.1016/j.clinthera.2011.03.003. PMID 21600388